CLINICAL TRIAL: NCT01873391
Title: Pain in Diagnostic Hysteroscopy: a Multivariate Analysis.
Brief Title: Pain in Diagnostic Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sandro Gerli (Other)
Responsible Party: Sponsor-Investigator, Sandro Gerli, Assistant Professor, Azienda Ospedaliera S. Maria della Misericordia
Organization: Azienda Ospedaliera S. Maria della Misericordia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: co2 vs h2o
Record Dates: First submitted 2013-06-01; First posted 2013-06-10 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Pain in Diagnostic Hysteroscopy
Keywords: Diagnostic hysteroscopy; Pain; VAS; Multivariate analysis; Normal saline; Carbon dioxide
MeSH Terms: conditions — Pain | interventions — Hysteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal saline (Active Comparator): Normal saline is a distension media of uterine cavity in diagnostic hysteroscopy.
  Interventions: Procedure: Diagnostic hysteroscopy
- Carbon dioxide (Active Comparator): Carbon dioxide is a distension media of uterine cavity in diagnostic hysteroscopy.
  Interventions: Procedure: Diagnostic hysteroscopy

INTERVENTIONS:
Procedure: Diagnostic hysteroscopy

SUMMARY:
The objective of this study is to assess which factors influence the pain perceived during diagnostic anesthesia-free hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* diagnostic hysteroscopy indication
* italian-speaking patients

Exclusion Criteria:

* patients who had previously undergone a diagnostic hysteroscopy
* patients who had been previously undergone to cervical surgery
* ongoing pregnancy
* cervical carcinoma
* pelvic inflammatory disease
* excessive uterine bleeding
* performance of an endometrial biopsy during the procedure

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain during diagnostic hysteroscopy by Visual Analogue Scale. | 5 minutes after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Gerli, MD, Study Director — University Of Perugia
Locations (1):
- Arbor Vitae Endoscopic Centre, Rome, Italy, Italy

REFERENCES:
- [Derived] Mazzon I, Favilli A, Grasso M, Horvath S, Bini V, Di Renzo GC, Gerli S. Pain in diagnostic hysteroscopy: a multivariate analysis after a randomized, controlled trial. Fertil Steril. 2014 Nov;102(5):1398-403. doi: 10.1016/j.fertnstert.2014.07.1249. Epub 2014 Sep 18. PMID 25241369